CLINICAL TRIAL: NCT01292252
Title: Assessment of the Efficacy of Forteo (Teriparatide) in Patients Undergoing Posterolateral Lumbar Spinal Fusion
Brief Title: Use of Forteo (Teriparatide) in Posterolateral Lumbar Spine Fusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shane Burch (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Shane Burch, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCSFSpineForteo
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Lumbar Spondylosis; Lumbar Spondylolisthesis; Adult Degenerative Lumbar Scoliosis
MeSH Terms: conditions — Spondylosis; Spondylolisthesis | interventions — Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Forteo, Terapeptide 20 ug subcutaneous injection
  Interventions: Biological: teriparatide
- Control (Placebo Comparator): Saline placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: teriparatide — Teriparatide 20 ug subcutaneous injection daily for 12 weeks
  Other Names: Forteo; recombinant human parathyroid hormone (1-34)
  Arms: Treatment
Biological: Placebo — Saline solution
  Arms: Control

SUMMARY:
The purpose of this study is to determine the effects of 12 weeks of daily treatment with teriparatide on spine fusion in adult patients who are undergoing multi-level posterolateral spine fusion surgery for degenerative conditions of the lumbar spine.

DETAILED DESCRIPTION:
For patients undergoing spine fusion surgery, non-fusion (or pseudarthrosis) is one of the major complications that can lead to poor clinical outcomes. Therefore, treatments that promote or augment fusion are highly desirable. Teriparatide (Forteo, recombinant human parathyroid hormone [1-34]) is a systemically administered peptide hormone that is FDA-approved for the treatment of osteoporosis in postmenopausal women or other populations at high risk for fracture. While teriparatide has been shown to enhance spinal fusion in several rodent and rabbit studies, no clinical studies to date have examined its effect on spinal fusion in humans. While Forteo is FDA approved, and IND is required for this trial to study an unapproved indication: Posterolateral Lumbar Spine Fusion.

This single-site two-year prospective randomized double-blind placebo-controlled study is designed to examine the effects of peri-operative teriparatide treatment in older adults undergoing multi-level posterolateral lumbar spine fusion. All eligible patients seen at the UCSF Spine Center will be invited to enroll in the study. Upon enrollment, patients will have screening labs drawn in conjunction with their routine pre-operative work-up, to include complete blood count (CBC), chemistry panel including calcium level, liver function tests (LFTs) including alkaline phosphatase, parathyroid hormone (PTH) level, and 25-hydroxyvitamin D level. If eligible after screening labs are completed, they will be scheduled for bone density (DEXA) scan and be randomized in a 2:1 ratio to receive daily subcutaneous injections of teriparatide 20 ug/d or placebo. The total duration of treatment will be 12 weeks, with two weeks pre-operative and 10 weeks post-operative treatment.

Patients will be scheduled to attend all standard post-operative follow-up clinic visits, which will be at 6 weeks, 3 months, 6 months, and 12 months after surgery. At 3 months post operative visit, patients will have lab drawn for calcium. At each follow-up visit, AP and lateral x-ray radiographs will be taken of the lumber spine to assess progression of bone healing and positioning of any hardware placed. Participants will be asked to complete a pain Visual Analog Score (VAS), European Quality of Life-5 Dimensions (EQ-5D), and Oswestry Disability Index (ODI) questionnaire at each visit for assessment of clinical outcomes. Thin-section helical CT scans of the lumbar spine will be taken at 12 months after surgery for definitive assessment of fusion. All radiographs will be evaluated by a blinded panel of three reviewers including a radiologist and a spine surgeon to assess primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60-90 years with lumbar spondylosis, spondylolithesis, or adult degenerative scoliosis, including disc pathology, stenosis, deformity, instability, or postdecompression revision, who are scheduled to undergo three-level or greater posterolateral lumbar spinal fusion.
* Willing and able to use a pen-type delivery system to administer daily subcutaneous injections.

Exclusion Criteria:

* Use of bone morphogenic protein (BMP) posterolaterally during the fusion procedure.
* Previous spinal fusion at the intended fusion levels.
* Prior use of Forteo (teriparatide).
* Use of digoxin.
* Paget's Disease of bone.
* History of primary skeletal malignancy, presence of bone metastases, or previous skeletal exposure to therapeutic irradiation.
* Elevated serum calcium, serum PTH >70 pg/ml, 25-hydroxyvitamin D <12 ng/mL, or active liver disease.
* History of symptomatic nephro- or urolithiasis in the past two years.
* History of malignant neoplasm in the past five years, except for superficial basal cell carcinoma or squamous cell carcinoma.
* Carcinoma in situ of the uterine cervix treated in the past year.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Burch, MD, Principal Investigator — University of California, San Francisco; Carmen Li, Study Director — University of California, San Francisco
Locations (1):
- UCSF Spine Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UCSF Spine Center — http://www.ucsfhealth.org/adult/medical_services/spine/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 714 patients were screened for the study between August 2011 and March 2016.
Groups:
- Treatment: Forteo, Terapeptide 20 ug: Forteo, Terapeptide 20 ug subcutaneous injection
  teriparatide: Teriparatide 20 ug subcutaneous injection daily for 12 weeks
- Control: Saline Placebo: Saline placebo
  Placebo: Saline solution
Period: Overall Study
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo
Started | 21 | 15
Completed | 21 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (6.1) | 71.3 (6.3) | 70.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 15 | 36
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (7.6) | 29.44 (6.4) | 28.48 (7.07)
Visual Analog Score (VAS) [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Score (VAS), the score range is 0-100 with higher scores indicating more pain
  units on a scale | 19.7 (9.6) | 15.2 (9.1) | 17.8 (9.5)
European Quality of Life - 5 Dimensions (EQ-5D) [Mean (Standard Deviation); unit: units on a scale] — European Quality of Life - 5 Dimensions (EQ-5D) is a standardized instrument for measuring generic health status, the scale range is from 0.000 (death) to 1.000 (perfect health)
  units on a scale | 0.57 (0.2) | 0.60 (0.2) | 0.58 (0.2)
Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index (ODI) provides information about how back or leg pain is affecting the ability to manage in everyday life, the points range from 0-50, which is doubled and reported as a percentage. Higher scores indicate higher disability.
  units on a scale | 52.1 (16.1) | 46.4 (15.3) | 49.7 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Spine Fusion, Measured by the Number of Participants With Complete Spine Fusion at 1 Year
Description: Quality of spine fusion, measured by the number of participants with complete spine fusion at 1 year. Spine fusion at one year was assessed using thin-section helical computed tomography (CT) scan of the lumbar spine.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo
Number analyzed (Participants) | 21 | 15
Participants | 11 | 6

2. Primary Outcome: Time to Spine Fusion
Time Frame: One year
Population: Data were not collected as intended and are not available to reported.
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Reported Outcomes Measured by: Visual Analog Score (VAS), European Quality of Life - 5 Dimensions (EQ-5D) and Oswestry Disability Index (ODI) Scores at 1 Year
Description: 1. The self-reported pain Visual Analog Score (VAS), the score range is 0-100 with higher scores indicating more pain.
  2. European Quality of Life - 5 Dimensions (EQ-5D) is a standardized instrument for measuring generic health status, the scale range is from 0.000 (death) to 1.000 (perfect health).
  3. Oswestry Disability Index (ODI) provides information about how back or leg pain is affecting the ability to manage in everyday life, the points range from 0-50, which is doubled and reported as a percentage. Higher scores indicate higher disability.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo
Number analyzed (Participants) | 21 | 15
units on a scale
  Visual Analog Score (VAS) | 11.67 (13.4) | 9.67 (8.0)
  European Quality of Life - 5 Dimensions (EQ-5D) | 0.733 (0.19) | 0.708 (0.17)
  Oswestry Disability Index (ODI) | 32.3 (19.9) | 31.9 (17.6)

4. Secondary Outcome: Adverse Effects
Description: Number of participants with serious adverse events and other (not including serious) adverse events at one year are reported.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo
Number analyzed (Participants) | 21 | 15
Participants
  Serious Adverse Events | 1 | 1
  Other (Not Including Serious) Adverse Events | 9 | 6

ADVERSE EVENTS:
Arm/Group | Treatment: Forteo, Terapeptide 20 ug | Control: Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/15
Other Adverse Events (participants affected / at risk) | 9/21 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Forteo, Terapeptide 20 ug (N=21) | Control: Saline Placebo (N=15)
myocardial infarction (Cardiac disorders) | 1 | 0
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Forteo, Terapeptide 20 ug (N=21) | Control: Saline Placebo (N=15)
constipation (Gastrointestinal disorders) | 2 | 1
dizziness (General disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 1 | 0
headache (General disorders) | 1 | 0
rapid heart (Cardiac disorders) | 1 | 0
skin rash (Skin and subcutaneous tissue disorders) | 1 | 0
insomnia (General disorders) | 1 | 0
chest pain (General disorders) | 1 | 0
infection of surgical site (Infections and infestations) | 1 | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
shingles (Infections and infestations) | 0 | 1
pain and burning at injection site (Skin and subcutaneous tissue disorders) | 0 | 3
altered mental state (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes